CLINICAL TRIAL: NCT05586048
Title: Effectiveness of Yiqi Fumai Lyophilized Injection for Acute Heart Failure: AUGUST-AHF Cohort Study
Brief Title: Effectiveness of Yiqi Fumai Lyophilized Injection for Acute Heart Failure
Acronym: AUGUST-AHF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Yan Liu, MD, Principal Investigator, China Academy of Chinese Medical Sciences
Other Study IDs: AUGUST-AHF cohort
Record Dates: First submitted 2022-10-13; First posted 2022-10-19 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Acute Heart Failure; Complementary Medicine; Chinese Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: patients who received YQFM
  Interventions: Drug: Yiqi Fumai Lyophilized Injection(YQFM)
- Non-exposed group: patients who didn't receive YQFM

INTERVENTIONS:
Drug: Yiqi Fumai Lyophilized Injection(YQFM) — No intervention was involved, but patients will be divided into exposed or non-exposed groups based on whether they received YQFM
  Groups: Exposed group

SUMMARY:
The goal of this cohort study is to observe the effectiveness of Yiqi Fumai Lyophilized Injection (YQFM) in patients with acute heart failure (AHF). It mainly aims to assess the effectiveness of YQFM on the 90-day mortality or readmission rate in patients with AHF and compare the results with AUGUST-AHF RCT study. There will be no intervention, but information will be collected during the hospital stay and during the follow-up period of 180 days . Researchers will compare exposed group(patients who received YQFM) and non-exposed group(patients who didn't received YQFM) to see if there is difference on the 90-day mortality or readmission rate.

DETAILED DESCRIPTION:
It mainly aims to assess the effectiveness of YQFM on the 90-day mortality or readmission rate in patients with AHF and compare the results with AUGUST-AHF RCT study. There will be no intervention, but patients will be asked to answer questions(such as scales or reporting of symptoms ) and provide biochemical or imaging tests, as well as undergo regular follow-up. Researchers will compare exposed group(patients who received YQFM) and non-exposed group(patients who didn't received YQFM) to see if there is difference on the 90-day mortality or readmission rate. We will also collect information on medication adherence during the follow-up period and remotely test patients during the follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AHF
* Age≥18 years
* Voluntarily participate in and sign the informed consent form

Exclusion Criteria:

* With major psychiatric disorders or unable to complete follow-up assessment
* Known allergies to drugs or drug ingredients
* Patients enrolled in other trials within 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AHF in China
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
90-day all-cause mortality or readmission for HF | 90-day
  90-day all-cause mortality or readmission for HF

SECONDARY OUTCOMES:
180-day all-cause mortality or HF readmission | 180-day
  180-day all-cause mortality or HF readmission
cardiac-specific death | 180 day
  cardiac-specific death
MACE | 180 day
  major cardiovascular adverse event
length of hospital stay | during the hospitalization of patients, an average of 10 days
  the length of patients staying in hospital
dyspnoea via visual analogue scale (VAS) | during the hospitalization of patients, an average of 10 days
  Dyspnea VAS scores range from a maximum of 10 to a minimum of 0. Higher scores mean a worse outcome. 10 means extreme dyspnea, and 0 means no dyspnea.
dyspnoea via Likert 7-point scale | during the hospitalization of patients, an average of 10 days
  The Likert 7-point scores range from a maximum of 7 to a minimum of 1. Higher scores mean a better outcome.
NYHA cardiac function classification | 180 day
  New York Heart Association cardiac function classification
Minnesota Living with Heart Failure Quality of Life (MLHFQ) scale | 180 day
  Likert 7-point scores range from a maximum of 105 to a minimum of 0. Higher scores mean a worse outcome.
Morisky Medication Adherence Scale (MMAS)-8 scale | 180 day
  MMAS-8 scores range from a maximum of 8 to a minimum of 0. Higher scores mean a better outcome
heart rate | 180 day
  heart rate
number of participants eligible for the randomized controlled trial of AUGUST-AHF | at admission
  Patients will complete a questionnaire with the help of researchers. This questionnaire includes the inclusion criteria for another study, the randomized controlled trial of AUGUST-AHF. After the patient has completed the questionnaire, the investigator will determine whether the patient meets the criteria based on the results

CONTACTS AND LOCATIONS:
Overall Officials: Xuecheng Zhang, MD, Study Director — Dongzhimen Hospital, Beijing
Locations (3):
- China (3):
  - Dongzhimen Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guizhou University of Traditional Chinese Medicine, Guiyang, Guiyang, Guizhou
  - The Second Affiliated Hospital of Guizhou University of Traditional Chinese Medicine, Guiyang, Guizhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang J, Sun Y, Zhou K, Zhang X, Chen Y, Hu J, Zhong C, Liu Y, Shang H. Rationale and design of the AUGUST-AHF Study. ESC Heart Fail. 2020 Oct;7(5):3124-3133. doi: 10.1002/ehf2.12787. Epub 2020 Jun 22. PMID 32567238
- [Derived] Zhang X, Kang J, Zhang J, Chen Y, Dai H, Hu M, Liu Y, Shang H. Effectiveness of Yiqi Fumai lyophilized injection for acute heart failure: Rationale and design of the AUGUST-AHF cohort study. Front Cardiovasc Med. 2023 Jan 10;9:1074406. doi: 10.3389/fcvm.2022.1074406. eCollection 2022. PMID 36704479